CLINICAL TRIAL: NCT06520449
Title: A Single-Arm Comparative Imaging Study of 68Ga-NTA-476 PET/CT Compared to Standard of Care 18F-DCFPyL PET/CT in Men With Prostate Cancer
Brief Title: 68Ga-NTA-476 Imaging in Prostate Cancer
Acronym: NTA-476
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Melbourne Theranostic Innovation Centre (Network)
Collaborators: 3B Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-07-851
Record Dates: First submitted 2024-07-21; First posted 2024-07-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; PET/CT; PSMA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-NTA-476 PET/CT Compared to Standard of Care 18F-DCFPyL PET/CT (Experimental): A single dose of 68Ga-NTA-476 will be administered on Day 1 of the study as an intravenous bolus injection under the supervision of the study Investigator or appropriately qualified delegate. The planned injected activity (IA) of 68Ga-NTA-476 is 2-3.5 MBq/kg.
  Following administration of 68Ga-NTA-476, participants will complete PET imaging at 0-30 minutes, 1 hour, and 4-6 hours. Each PET scan will take up to 30 minutes.
  Interventions: Drug: 68Ga-NTA-476

INTERVENTIONS:
Drug: 68Ga-NTA-476 — The novel Prostate Specific Membrane Antigen (PSMA) targeting molecule, NTA-476, is comprised of a small peptide targeting moiety that is attached to a linker and dodecane tetraacetic acid (DOTA) cage which enables chelation of the radionuclide 68Ga for Positron Emission Tomography (PET) imaging.

SUMMARY:
This study is investigating a new agent to be used in PET imaging for prostate cancer, called 68Ga-NTA-476. It aims to find out where 68Ga-NTA-476 goes in the body once it is injected into a person and whether there are any side effects or issues with tolerating the compound. This will be compared to an existing imaging compound which is currently used in Australia called 18F-DCFPyl. 68Ga-NTA-476 has been developed and tested in the laboratory; however, this is the first time that it will be tested in humans.

DETAILED DESCRIPTION:
This study is investigating a new agent to be used in PET imaging for prostate cancer, called 68Ga-NTA-476. It aims to find out where 68Ga-NTA-476 goes in the body once it is injected into a person and whether there are any side effects or issues with tolerating the compound. This will be compared to an existing imaging compound which is currently used in Australia called 18F-DCFPyl. 68Ga-NTA-476 has been developed and tested in the laboratory; however, this is the first time that it will be tested in humans.

Who is it for? You may be eligible for this study if you are an adult older than 18 years of age, you have been diagnosed with prostate cancer and do not have any significant other health issues.

Study details All participants who choose to participate will complete a Screening Visit to make sure that they meet the eligibility requirements for the study. Procedures completed during this visit will include demographic details, medical history, physical examination, vital signs, ECG, blood samples to check overall health status and a 18F-DCFPyl PET scan.

Following confirmation of eligibility, participants will complete an Imaging Day Visit. During this visit, single dose of 68Ga-NTA-476 will be injected via a vein into the body. Following this, PET scans will be completed at about 0-30 minutes, 1 hour, and 4-6 hours. Participants will be observed in the clinical for a total of 6 hours to check vital signs and record any side effects.

Between 7-9 days after this, a final study visit will be completed. Blood samples will be collected to check overall health status and the research team will check to see if any side effects were experienced.

A total of 10 participants will be enrolled in this study at Melbourne Theranostic Innovation Centre in Australia

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent prior to start of any study procedures and assessments and must be willing to comply with all study procedures.
2. Adult participants = 18 years of age.
3. Participants with a documented history of histologically confirmed diagnosis of prostate cancer.

   * Participants must have PSA > 0.1 ng/mL.
   * Participants on chemotherapy may be approved on a case-by-case basis at the principal investigator's discretion if the last dose of chemotherapy is administered at least 3 weeks prior to receipt of 68Ga-NTA-476, and subsequent dose of chemotherapy are to resume following completion of End of Treatment Visit (EOTV), if it is determined not to put the patient at an increased risk of adverse drug effects and/or interfere with the integrity of study outcome.
   * Participants on other anti-cancer therapy, such as novel anti-androgen therapy, may be allowed on a case-by-case basis at the principal investigator's discretion, with an agreement of a washout period prior to 68Ga-NTA-476 dosing, if it is determined not to put the patient at an increased risk of adverse drug effects and/or interfere with the integrity of study outcome.
4. Eastern Cooperative Oncology Group (ECOG) performance status = 2.
5. Participants must have a life expectancy of >3 months in the opinion of the Investigator.
6. Male participants who are able to father a child must agree to avoid impregnating a partner and to adhere to a highly effective method of contraception during the study and for 14 days after the last injection of 68Ga-NTA-476. Participants must agree to not donate sperm during the study and for 14 days after the injection of 68Ga-NTA-476. Acceptable methods of contraception are described in section 14.3.1 of the Protocol.

   Exclusion Criteria:
7. Have any medical condition that would, in the Investigator's judgment, prevent the participant's full participation in the clinical study due to safety concerns or compliance with clinical study procedures, including but not limited to participants with severe claustrophobia.
8. Residual toxicity > Grade 1 from prior/current anti-cancer therapy (except alopecia). Participants with > Grade 1 toxicity from prior anti-cancer therapy may be approved on a case-by-case basis at the principal investigator's discretion, if it is determined not to put the patient at an increased risk of adverse drug effects and/or interfere with the integrity of study outcome.
9. History of uncontrolled allergic reactions and/or known or expected hypersensitivity to peptide therapeutics, including 68Ga-NTA-476 or any of its excipients.
10. Inadequate organ functions as reflected in laboratory parameters:

    * Creatinine clearance (calculated using Cockcroft-Gault formula, or measured) < 60 mL/min or serum creatinine >1.5 x upper limit of normal (ULN)
    * Platelet count of < 75 x 109/L
    * Absolute neutrophil count (ANC) < 1.0 x 109/L
    * Haemoglobin < 9 g/dL
    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 x ULN, or > 5 x ULN for patients with known liver metastases
    * Total bilirubin > 1.5 x ULN, except for patients with documented Gilbert's syndrome who are eligible if total bilirubin = 3 x ULN
11. For participants not taking warfarin or other anticoagulants: international normalised ratio (INR) =1.5 or prothrombin time (PT) =1.5 x ULN; and either partial thromboplastin time or activated partial thromboplastin time (PTT or aPTT) =1.5 x ULN. Participants taking warfarin must be on a stable dose that results in a stable INR <3.5. Among participants receiving other anticoagulant therapy, PT or aPTT must be within the intended therapeutic range of the anticoagulant.
12. Major surgery within 28 days prior to the dose of 68Ga-NTA-476. Exceptions may be approved on a case-by-case basis at the principal investigator's discretion, if it is determined not to put the participant at an increased risk of adverse drug effects and/or interfere with the integrity of study outcome.
13. Any uncontrolled intercurrent illness or clinically significant uncontrolled condition(s), including but not limited to active bacterial, fungal, or viral infections requiring systemic therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — For men with prostate cancer
Enrollment: 10 (Actual)
Dates: Start 2024-09-13 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Tumour uptake of 68Ga-NTA-476 as compared to 15F-DCFPyl in participants with prostate cancer | PET/CT scans completed at 0-30 minutes, 1 hour, and 4-6 hours following 68Ga-NTA-476 administration
  Standardised Uptake Value (SUV)max, SUVmean and total tumour volume by PET/CT quantitation
To characterize the uptake and washout of 68Ga-NTA-476 in normal organs as compared to 18F-DCFPyL in participants with prostate cancer | PET/CT scans completed at 0-30 minutes, 1 hour, and 4-6 hours following 68Ga-NTA-476 administration
  Time Activity Curves (TACs), describing % of the injected activity vs time will be derived for selected organs and tumours

SECONDARY OUTCOMES:
To assess the safety and tolerability of a single dose of 68Ga-NTA-476 | Safety will be assessed on the Imaging Day in the clinic during observation for up to 6 hours post injection of 68Ga-NTA-476 and followed up for a total of 1 week following administration.
  Safety is evaluated with the properties, incidence, nature and severity of AEs and SAEs, abnormal laboratory parameters, vital signs, and electrocardiogram (ECG) results per Common Terminology Criteria for Adverse Events (CTCAE) v5.0
To explore the dosimetry of 68Ga-NTA-476 | PET/CT scans completed at 0-30 minutes, 1 hour, and 4-6 hours following 68Ga-NTA-476 administration
  Absorbed radiation doses of 68Ga-NTA-476 in critical organs (e.g., kidneys, bone marrow)

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Rod Hicks, MB BS, MD, FRACP, FICIS, Principal Investigator — Melbourne Theranostic Innovation Centre
Locations (1):
- Melbourne Theranostic Innovation Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
PICF does not allow for sharing of IPD